CLINICAL TRIAL: NCT00833729
Title: An Open Label, Prospective Cohort Pilot Study to Evaluate the Efficacy and Safety of Etanercept in the Treatment of Moderate to Severe Plaque Psoriasis in Patients Who Have Not Had an Adequate Response to Adalimumab
Brief Title: The Safety & Efficacy of Etanercept in Psoriasis Patients Who Have Not Responded to Adalimumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatrials Research (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Ronald Vender MD FRCPC, Principal Investigator, Dermatrials Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-2008-0008
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis; etanercept; adalimumab; moderate to severe plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

ARMS (1):
- etanercept (Experimental): Single armed study
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — 50 mg twice weekly (BIW) for 12 wks followed by a dose reduction to 50mg once weekly (OW) for an additional 12 weeks.

SUMMARY:
To describe the response of etanercept after adalimumab has failed to produce a satisfactory response in moderate to severe plaque psoriasis. A total of 10 patients with moderate to severe psoriasis who are currently using adalimumab for at least 12 weeks but have a PGA of mild or worse will be transitioned to etanercept 50 mg twice weekly (BIW) for 12 wks followed by a dose reduction to 50mg once weekly (OW) for an additional 12 weeks.

DETAILED DESCRIPTION:
A total of 10 patients with moderate to severe psoriasis who are currently using adalimumab for at least 12 weeks but have a PGA of mild or worse will be transitioned to etanercept 50 mg twice weekly (BIW) for 12 wks followed by a dose reduction to 50mg once weekly (OW) for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject has had a diagnosis of moderate to severe chronic plaque psoriasis for at least 6 months
* Subject has had a sub-optimal response to continuous treatment with adalimumab administered for at least 3 consecutive months prior to screening, with no treatment interruptions exceeding 14 days, at doses of 40 mg every other week (eow) after a loading of 80mg sc. The last dose of adalimumab must be greater than 11 days and less than 17 days before the first dose of etanercept.
* PGA of mild or worse
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile or is of childbearing potential and is practicing an approved method of birth control throughout the study. The results of a urine pregnancy test performed at the screening visit must be negative.
* Subject is judged to be in generally good health as determined by the Investigator based upon the results of medical history, laboratory profile, and physical examination performed at screening.
* Subject must be able to self-administer or has a qualified designee who can reliably administer SC injections.
* Subject must be able and willing to give written informed consent and to comply with the requirements of this study protocol.
* Subject has a negative PPD test at within 6 months of screening.
* Able to start etanercept per the approved Enbrel® product monograph

Exclusion Criteria:

* Previous treatment with etanercept
* Subject receives or requires:
* UVB phototherapy, (other than narrow-band UVB), excessive sun exposure or the use of tanning booths within 14 days prior to Baseline visit.
* PUVA phototherapy within 14 days prior to Baseline visit.
* Systemic non-biologic therapies for psoriasis within 30 days prior to Baseline visit.
* Biologic therapies (excluding adalimumab) for psoriasis within 30 days prior to Baseline visit.
* High potentcy topical steroids during the study period
* Received any investigational agent within 30 days or 5 half lives prior to Baseline (whichever is longer), or within a duration of its known pharmacological activity.
* Subject has other active skin diseases or skin infections (bacterial, fungal, viral or parasitic) that may interfere with evaluation of psoriasis.
* Infection(s) requiring treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to Baseline or oral antibiotics, oral antivirals, or oral antifungals within 14 days prior to Baseline.
* History of moderate to severe congestive heart failure (NYHA class III or IV), recent cerebrovascular accident and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
* History of CNS demyelinating disease or neurologic symptoms suggestive of CNS demyelinating disease.
* History of listeriosis, histoplasmosis, chronic or active Hepatitis B infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active TB.
* Known hypersensitivity to the excipients of etanercept as stated in the label.
* Erythrodermic psoriasis generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis or new onset guttate psoriasis.
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.
* History of clinically significant drug or alcohol abuse in the last 12 months.
* Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study and not able to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Mean change in PGA score | Baseline to 12 weeks

SECONDARY OUTCOMES:
Mean change in body surface area covered in psoriasis | Baseline to 12 weeks and again at 24 weeks
Mean change in DLQI | Baseline to 12 weeks and again at 24 weeks
Treatment satisfaction | Baseline to 12 weeks and again at 24 weeks
Proportion of patients achieving an improvement in PGA score | Baseline to 12 weeks and again at 24 weeks
Mean change in adverse events | Baseline to 12 weeks and again at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Vender, MD FRCPC, Principal Investigator — Dermatrials Research
Locations (1):
- Dermatrials Research, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Vender R. An open-label, prospective cohort pilot study to evaluate the efficacy and safety of etanercept in the treatment of moderate to severe plaque psoriasis in patients who have not had an adequate response to adalimumab. J Drugs Dermatol. 2011 Apr;10(4):396-402. PMID 21455550